CLINICAL TRIAL: NCT01460628
Title: The Effect of Armodafinil (Nuvigil) on Fatigue and Quality of Life in Peri- and Postmenopausal Women
Brief Title: Effect of Nuvigil on Fatigue
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Hadine Joffe, MD, Vice Chair for Research, Psychiatry Department, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011P-001055
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Menopause
Keywords: fatigue; menopausal symptoms; hot flashes; Vasomotor symptoms; perimenopause; related Quality of life
MeSH Terms: conditions — Fatigue; Hot Flashes | interventions — Modafinil

ARMS (1):
- Armodafinil (Experimental): Armodafinil is the drug being tested.
  Interventions: Drug: Armodafinil

INTERVENTIONS:
Drug: Armodafinil — Women who are eligible will receive 4 weeks of treatment with armodafinil. Armodafinil will be titrated from 50-mg/day up to 150-mg/day. For exploratory reasons only, at the end of the 4-week treatment period, participants will enter a discontinuation phase in which they will be randomized to double-blind treatment with armodafinil 150-mg/day or matching placebo for 2 weeks in a 1-to-1 ratio. No primary outcomes were studied in the discontinuation phase.
  Other Names: Nuvigil

SUMMARY:
The purpose of this study is to determine if armodafinil improves quality of life and is an effective treatment of fatigue in symptomatic perimenopausal and postmenopausal women.

DETAILED DESCRIPTION:
Fatigue is one of the most prevalent symptoms occurring in peri- and postmenopausal women. It is strongly associated with reduced quality of life in this population. Studies have shown a strong association between fatigue and menopausal symptoms such as hot flashes, vaginal symptoms, and sexual dysfunction. Because sleep disturbance commonly co-occurs in women with hot flashes as a result of nocturnal hot flashes disrupting sleep, sleep disturbance may explain the association between hot flashes and fatigue in this population. However evidence suggests that fatigue can occur in the absence of sleep disruption, indicating that sleep problems do not exclusively explain the etiology of fatigue in this population.

Armodafinil is a wakefulness-promoting agent that acts as a central nervous system stimulant. It is chemically and pharmacologically unrelated to other CNS stimulants, such as methylphenidate and amphetamine. Armodafinil is FDA approved to increase wakefulness in patients with excessive sleepiness due to narcolepsy, obstructive sleep apnea, and shift work sleep disorder. It has not be studied in menopause-associated fatigue.

In the proposed study, the investigators plan to investigate the effect of armodafinil on quality of life and fatigue in a population of peri- and postmenopausal women with fatigue and reduced quality of life who do not have primary sleep disorders, significant levels of insomnia, or depression.

ELIGIBILITY:
Inclusion Criteria:

Women

* Ages 40-65
* Peri- and postmenopausal
* Suffering from fatigue
* Experiencing hot flashes(Not required for perimenopausal women)

Exclusion Criteria:

* Current episode of major depression
* Moderate-to-severe insomnia
* Night shift workers
* Previous diagnosis of manic depressive disorder, psychotic disorder, or psychotic symptoms
* Suicidal ideation
* Alcohol/drug abuse
* Concern about potential misuse of study medication
* Use of prescribed medications to treat insomnia or other sleep disturbance symptoms
* Pregnant or breastfeeding
* Use of systemic menopausal hormonal therapy or birth control
* Use of centrally active medications, such as antidepressants, anxiolytics, and hypnotics agents
* Use of clopidogrel
* Use of atomoxetine
* Cardiovascular contraindications of use of armodafinil

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadine Joffe, MD, MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Armodafinil: Armodafinil is the drug being tested. Women who are eligible will receive 4 weeks of treatment with armodafinil. Armodafinil will be titrated from 50-mg/day up to 150-mg/day. For exploratory reasons only, at the end of the 4-week treatment period, participants will enter a discontinuation phase in which they will be randomized to double-blind treatment with armodafinil 150-mg/day or matching placebo for 2 weeks in a 1-to-1 ratio.
Period: Overall Study
Arm/Group | Armodafinil
Started | 25
Completed | 20
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Armodafinil
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (5.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Menopause Quality Of Life Questionnaire (MENQOL) Physical Domain Subscale
Description: This is a widely used self-report instrument to determine differences in quality of life among menopausal women and to measure changes in their quality of life over time. Four domain scores are calculated from the 29-item instrument. The physical domain subscale has 16 questions and a range from 0-8 with higher scores indicating worse symptoms.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Armodafinil
Number analyzed (Participants) | 20
units on a scale | 1.9 [1.3 to 2.7]

2. Primary Outcome: Brief Fatigue Inventory (BFI)
Description: This is a widely used self-report instrument to assess the severity of fatigue and the impact of fatigue on daily functioning. This 9 item instrument yields a global fatigue score ranging from 0-10 with higher scores indicating worse symptoms. .
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Armodafinil
Number analyzed (Participants) | 20
units on a scale | 2.2 [1.1 to 4.4]

3. Secondary Outcome: Epsworth Sleepiness Scale (ESS)
Description: This self-report scale is widely used as a subjective measure of sleepiness. This 8 item instrument yields a total score ranging from 0-24 with higher scores indicating worse symptoms.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Armodafinil
Number analyzed (Participants) | 20
units on a scale | 3.0 [1.0 to 5.5]

4. Secondary Outcome: Hot Flash Frequency (24-hr Period)
Description: The Daily Vasomotor Symptom Diary consists of a 7-day scale on which the subject records the total number of hot flushes they experience on a daily basis. Weekly averages for a 24-hour period are calculated.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: # of hot flashes
Arm/Group | Armodafinil
Number analyzed (Participants) | 20
# of hot flashes | 1.5 [0.4 to 2.4]

5. Secondary Outcome: Symptom Checklist-10 Anxiety
Description: The SCL-10 anxiety subscale, developed from the refinement of the Hopkins Symptom Checklist (HSCL), consists of 10 questions focused on how much discomfort symptoms of anxiety (e.g. "nervousness or shaking inside") have caused in the past two weeks. Each question is answered on a scale from 0-4, and answers are averaged for a total score between 0-4 with higher scores indicating more anxiety.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Armodafinil
Number analyzed (Participants) | 20
units on a scale | 0 [0 to 0.2]

6. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 is the self-administered form of the Primary Care Evaluation of Mental Disorders (PRIME-MD), a widely used instrument designed to screen for psychiatric illnesses in primary-care settings. This 9-item instrument assesses mood, depressive symptoms, and suicidal ideation. The range of total scores is 0-27 with higher scores indicating worse symptoms. Generally, scores 5-9 indicate mild depression, 10-14 indicate moderate depression, and 15+ indicate moderately severe or severe depression.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Armodafinil
Number analyzed (Participants) | 20
units on a scale | 3.0 [1.0 to 6.0]

7. Secondary Outcome: Brown Attention Deficit Disorder Scale (BADDS)
Description: This is a normed and validated measure of ADHD-related executive function impairments. The clinician administered scale measures five clusters of executive function including 1) organizing and activating for work, 2) sustaining attention and concentration, 3) sustaining alertness, effort, and processing speed, 4) managing affective interference, and 5) using working memory and accessing recall. The frequency and severity of each of the 40 items is rated on a scale of 0 to 3, with the total scores ranging from 0-120 and higher scores indicating worse symptoms.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Armodafinil
Number analyzed (Participants) | 20
units on a scale | 15.5 [5.5 to 25]

ADVERSE EVENTS:
Arm/Group | Armodafinil
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 16/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil (N=25)
headache (Nervous system disorders) | 3 (3)
increased blood pressure or heartbeat (Cardiac disorders) | 4 (4)
dry mouth (Ear and labyrinth disorders) | 3 (4)
jaw clenching (Musculoskeletal and connective tissue disorders) | 1 (2)
stomach ache/nausea/gas (Gastrointestinal disorders) | 7 (9)
upper respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 5 (7)
sleep disruption (Nervous system disorders) | 4 (5)
depression/anxiety (Psychiatric disorders) | 8 (9)
dizziness (Ear and labyrinth disorders) | 1 (1)
jitteriness (Nervous system disorders) | 1 (1)
constipation/diarrhea (Gastrointestinal disorders) | 4 (4)
skin irritation (Skin and subcutaneous tissue disorders) | 3 (3)
increased appetite (Metabolism and nutrition disorders) | 1 (1)
spotting (Reproductive system and breast disorders) | 1 (1)
word recall (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No